CLINICAL TRIAL: NCT01687686
Title: Differential Effects of Total Cholesterol, Non-HDL Cholesterol and Triglycerides on Initial Presentation of Specific Cardiovascular Diseases (a CALIBER Study)
Brief Title: Differential Effects of Lipids on Cardiovascular Diseases: A CALIBER Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Owen Nicholas, Senior Medical Statistician, University College, London
Other Study IDs: CALIBER-12-01
Record Dates: First submitted 2012-09-13; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Stable Angina; Unstable Angina; Non ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction; Myocardial Infarction Not Otherwise Specified
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All cohort: Initially healthy patients in General Practise Research Database (GPRD) meeting the inclusion criteria at any point between 1st January 2001 and 25th March 2010

SUMMARY:
The role of lipids as risk factors for cardiovascular events is well-documented, although events studied have largely been broad classes without specific detail. This study will examine a more refined set of endpoints.

DETAILED DESCRIPTION:
The role of lipids (cholesterol and triglycerides) as risk factors for cardiovascular events is well-documented. The Emerging Risk Factors Collaboration found approximately log-linear adjusted associations of cholesterol concentrations with risks of first-time non-fatal myocardial infarction; coronary heart disease (CHD) death; ischaemic, haemorrhagic and unclassified stroke. They also found that triglycerides concentration was not independently related with CHD risk after controlling for HDL cholesterol (HDL-C), non-HDL-C, and other standard risk factors. The Prospective Studies Collaboration found that Higher HDL-C and lower non-HDL-C levels were approximately independently associated with lower ischaemic heart disease mortality. By focusing on broad outcomes these large meta-analyses conflate the association between development of the different cardiovascular disease (CVD) phenotypes, disease progression and mortality from cardiovascular causes.

With linked electronic health records, we have the potential for a cohort with sufficient size and clinical detail to investigate the association between lipid concentrations and initial presentation of a range of CVD phenotypes across cerebral, coronary, abdominal and peripheral arterial circulations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 100, had at least one year of electronic health record data which meet General Practice Research Database data quality standards

Exclusion Criteria:

* No record indicating any cardiovascular disease phenotypes

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort used in the present analysis was drawn from patients registered with 225 GPRD general practices in England which consented to data linkage, covering approximately 5% of the UK population. We used an open cohort design, where participants joined the cohort when they met the inclusion criteria at any point between 1st January 2001 and 25th March 2010, the date of the last GPRD data submission. Patients were included in cohort if, prior to study entry, they were aged 30 to 100, had at least one year of electronic health record data which meet General Practice Research Database data quality standards, and had no record indicating any cardiovascular disease phenotypes. Patients were followed up until the date of an initial presentation of one of our cardiovascular endpoints or were censored on the date of leaving the practice or the date of last data submission from their practice.
Sampling Method: Non-Probability Sample
Enrollment: 175872 (Actual)
Dates: Start 2001-01; Primary Completion 2010-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Rate of stable angina | Cohort followed up for average of 7 years
  Incidence of stable angina in study population

SECONDARY OUTCOMES:
Rate of unstable angina | Cohort followed up for average of 7 years
  Incidence of unstable angina in study population

OTHER OUTCOMES:
Rate of non ST elevation myocardial infarction | Cohort followed up for average of 7 years
  Incidence of non ST elevation myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, Greater London, United Kingdom

REFERENCES:
- [Background] Prospective Studies Collaboration; Lewington S, Whitlock G, Clarke R, Sherliker P, Emberson J, Halsey J, Qizilbash N, Peto R, Collins R. Blood cholesterol and vascular mortality by age, sex, and blood pressure: a meta-analysis of individual data from 61 prospective studies with 55,000 vascular deaths. Lancet. 2007 Dec 1;370(9602):1829-39. doi: 10.1016/S0140-6736(07)61778-4. PMID 18061058
- [Background] Emerging Risk Factors Collaboration; Di Angelantonio E, Sarwar N, Perry P, Kaptoge S, Ray KK, Thompson A, Wood AM, Lewington S, Sattar N, Packard CJ, Collins R, Thompson SG, Danesh J. Major lipids, apolipoproteins, and risk of vascular disease. JAMA. 2009 Nov 11;302(18):1993-2000. doi: 10.1001/jama.2009.1619. PMID 19903920
- [Background] Ebrahim S, Sung J, Song YM, Ferrer RL, Lawlor DA, Davey Smith G. Serum cholesterol, haemorrhagic stroke, ischaemic stroke, and myocardial infarction: Korean national health system prospective cohort study. BMJ. 2006 Jul 1;333(7557):22. doi: 10.1136/bmj.38855.610324.80. Epub 2006 Jun 6. PMID 16757495